CLINICAL TRIAL: NCT05013892
Title: Phase II Trial of Normal Tissue Sparing Whole Brain Radiation Therapy (NTS-WBRT) in Patients With Brain Metastases
Brief Title: NTS-WBRT in Brain Metastases
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Helen A. Shih, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-356
Record Dates: First submitted 2021-08-06; First posted 2021-08-19 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Brain Metastases
Keywords: Brain Metastases
MeSH Terms: conditions — Brain Neoplasms | interventions — Radiotherapy; Memantine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- NTS-WBRT (normal tissue sparing whole brain radiation therapy) + Memantine (Experimental): Participants will be randomly assigned to NTS-WBRT (normal tissue sparing whole brain radiation therapy) administration group and receive:
  * NTS-WBRT for 5 days (Monday-Friday) for either 2 or 3 weeks.
  * Memantine per standard of care, 1-2x daily for up to 24 weeks Specific participant administration schedules will be determined by study doctor
  Interventions: Radiation: NTS-WBRT (normal tissue sparing whole brain radiation therapy); Drug: Memantine

INTERVENTIONS:
Radiation: NTS-WBRT (normal tissue sparing whole brain radiation therapy) — Radiation
  Other Names: Radiation Therapy
Drug: Memantine — Capsule, taken orally
  Other Names: Namenda; Namenda XR; Namenda XR Titration Pack

SUMMARY:
This research is being done to assess the quality of life and symptom burden in participants who receive (normal tissue sparing whole brain radiation therapy (NTS-WBRT).

This research study involves:

* NTS-WBRT (normal tissue sparing whole brain radiation therapy)
* Memantine standard of care drug

DETAILED DESCRIPTION:
This is a Phase 2 trial testing the safety and effectiveness of NTS-WBRT (normal tissue sparing whole brain radiation therapy) in treating brain metastases.

NTS-WBRT is a targeted radiation therapy that further reduces radiation dose to tissue that does not need radiation therapy treatment.

The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.

It is expected that about 41 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with a solid tumor diagnosis and any number of brain metastasis clinically indicated for cranial irradiation with whole brain radiation therapy
* Age ≥ 18
* Karnofsky Performance Status ≥ 70
* Prior stereotactic radiosurgery (SRS) permissible per physician discretion
* Prior craniotomy permissible per physician discretion. Protocol radiation therapy should be initiated ≥2 weeks after craniotomy.
* Prior partial brain radiation therapy permissible if target volume < 50% brain and per physician discretion
* Expectant > 6 months survival
* Ability to understand and the willingness to sign a written informed consent document.
* Fluency in English, able to complete questionnaires and neurocognitive testing
* Ability to undergo MRI with gadolinium examination
* Ability to return for follow-up examinations throughout the course of this study for a maximum of 2 years after radiation treatment completion
* Any prior, concomitant, or post-radiotherapy systemic therapy is permitted at discretion of treating physicians
* Negative pregnancy test for premenopausal women

Exclusion Criteria:

* Leptomeningeal disease (by any one or more of clinical assessment, radiographic assessment, or cerebrospinal fluid study)
* Prior whole brain radiation therapy
* Pre-existing or current use of memantine or other NMDA antagonists
* Known allergy to contrast used in imaging studies and/or inability to have MRI imaging
* Uncontrolled intercurrent illness that could significantly affect baseline cognitive function as determined by the enrolling clinician, such as symptomatic congestive heart failure, unstable angina pectoris, prior CVA, significant uncontrolled epilepsy or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or unwilling to use appropriate contraception to prevent pregnancy during the time of radiation therapy
* Concurrent participation in an investigational systemic therapy protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2022-02-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Patient Reported Quality of Life for NTS-WBRT (normal tissue sparing whole brain radiation therapy) | 4 Months
  Assessed by Functional Assessment of Cancer Therapy-Brain (FACT-Br) questionnaire. Score range is 0-200 and the higher the score, the better the outcome.
Change in Patient Reported Symptom Burden for NTS-WBRT (normal tissue sparing whole brain radiation therapy) | 4 Months
  Assessed by Functional Assessment of Cancer Therapy-Brain (FACT-Br) questionnaire. Score range is 0-200 and the higher the score, the better the outcome.

SECONDARY OUTCOMES:
Tumor local control Rates between NTS-WBRT+SIB and NTS-WBRT | baseline, 2, 4, 6, 9, 12, 18 and 24 months
  Estimated by the cumulative incidence function treating death as a competing risk, compared using Gray's test
Intracranial- Progression Free Survival (PFS) between NTS-WBRT+SIB and NTS-WBRT | baseline, 2, 4, 6, 9, 12, 18 and 24 months
  Estimated using the Kaplan-Meier method, compared using the logrank test
Overall survival (OS) between NTS-WBRT+SIB and NTS-WBRT | The date of randomization to the date of death, or otherwise censored at the last follow-up date for patients still alive up to 24 months
  Estimated using the Kaplan-Meier method, compared using the logrank test
Change in Neurocognitive function between NTS-WBRT+SIB and NTS-WBRT | baseline, 2, 4, 6, 9, 12, 18 and 24 months
  Assessed longitudinally by the HADS-D and HADS-A questionnaires
Change in Mood between NTS-WBRT+SIB and NTS-WBRT | baseline, 2, 4, 6, 9, 12, 18 and 24 months
  Mixed effects models with treatment arm as a fixed effect will be used to compare changes in depression (HADS-D) and anxiety (HADS-A) scores over time
Change in Fatigue between NTS-WBRT+SIB and NTS-WBRT | baseline, 2, 4, 6, 9, 12, 18 and 24 months
  Mixed effects models with treatment arm as a fixed effect will be used to compare changes in the fatigue score over time
Change in Neuroendocrine function between NTS-WBRT+SIB and NTS-WBRT | baseline, 2, 4, 6, 9, 12, 18 and 24 months
  Estimated by the cumulative incidence function treating intracranial progression and death as competing risks; compared using Gray's test.
Change in Hearing between NTS-WBRT+SIB and NTS-WBRT Assessed by Pure Tone Average | baseline, 2, 4, 6, 9, 12, 18 and 24 months
  Changes in pure tone average (PTA) from baseline to each subsequent assessment will be compared between treatment arms using Wilcox rank-sum test. Pure tone thresholds are found by presenting tones using standard headphones and methods in a sound treated booth. Pure tone thresholds will be tested by both bone (500, 1000, 2000 and 4000 Hz) and air conduction (250, 500, 1000, 2000, 3000, 4000, 6000, 8000, 10000, 12000, and 14000 Hz). Masking will be applied sufficient to determine the ear responsible for each value. The results of this testing will be used to determine the sensorineural hearing level. If significant conductive loss is found, bone conduction threshold will be used to report sensory ototoxicity. Threshold effects across frequency will be combined into a Pure Tone Average (PTA), defined as the average of audiometric thresholds at 500, 1000, 2000, and 4000. A significant decrease in Pure Tone Average is defined as an increase > 10 dB in relation to baseline threshold.
Change in Hearing between NTS-WBRT+SIB and NTS-WBRT Assessed by Word Recognition Score | baseline, 2, 4, 6, 9, 12, 18 and 24 months
  Changes in word recognition score (WRS) from baseline to each subsequent assessment will be compared between treatment arms using Wilcox rank-sum test. Word recognition is defined as the percent correct on a standard, 50-item word list of English monosyllables: CID W-22, NU#6 or CNC. A significant decrease in word recognition is defined as a score exceeding the 95% critical difference from the table of Thornton and Raffin.
Change in Hearing between NTS-WBRT+SIB and NTS-WBRT Assessed by Otoacoustic Emissions | baseline, 2, 4, 6, 9, 12, 18 and 24 months
  The rates of absent otoacoustic emissions (OAE) will be compared between treatment arms using Fisher's exact test. The OAE (Otoacoustic Emissions) test checks part of the inner ear's response to sound. Otoacoustic emissions are sounds given off by one small part of the cochlea when it is stimulated by soft clicking sounds. When the sound stimulates the cochlea, the outer hair cells vibrate. The vibration produces a nearly inaudible sound that echoes back into the middle ear. The results are either present or absent. Present OAEs are consistent with normal to near normal hearing. Absent OAEs may be a sign of a problem related to study treatment.
Alopecia Rates between NTS-WBRT+SIB and NTS-WBRT | baseline, 2, 4, 6, 9, 12, 18 and 24 months
  Assessed by patient report and visual inspection with documented photography; compared by Fisher's exact test
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE Version 5.0 | Up to 24 months
  The number and proportion of adverse events, graded as defined by CTCAE version 5.0 will be tabulated by type and grade, compared using Fisher's exact test.

CONTACTS AND LOCATIONS:
Overall Officials: Helen A Shih, MD, MS, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation